CLINICAL TRIAL: NCT01101750
Title: Immunogenicity Of A Prophylactic Quadrivalent Human Papillomavirus (Types 6, 11, 16, And 18) L1 Virus-Like Particle Vaccine In Male And Female Adolescent Transplant Recipients.
Brief Title: Does the HPV Vaccine Cause the Same Response in Adolescent Kidney and Liver Transplant Patients as in Healthy Controls?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GardasilMerckGomez-Lobo
Record Dates: First submitted 2010-04-05; First posted 2010-04-12 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Cervical Cancer; Hpv; Warts
Keywords: Gardasil; HPV; transplant; adolescent; prevention; vaccine; immunogenicity; vaccination
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; Warts | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Intervention Model Description: Prospective study to evaluate immune response to the Gardisil vaccine in patients with a history of liver transplant and patients with a history of kidney transplant.
Masking Description: No masking.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liver and Kidney Transplant Patient Arm (Other): Standard of Care Intervention: Participants on this arm receive Gardasil vaccine and have a history of liver or kidney transplant.
  Interventions: Biological: Quadrivalent HPV for types 6, 11, 16 and 18

INTERVENTIONS:
Biological: Quadrivalent HPV for types 6, 11, 16 and 18 — Per standard of care, Gardasil 0.5ml IM injection on day one, month 2, and month 6.
  Serum samples on day one, month 3 and month 7.
  Other Names: Gardasil Vaccine

SUMMARY:
The purpose of the study is to understand if children with liver and kidney transplants develop the antibodies from the Gardasil vaccine.

The Gardasil vaccine protects against Human Papilloma Virus (HPV) types 16 and 18, which cause most types of cancers of the cervix, vagina and vulva. It also protects against Human Papilloma Virus types 6 and 11, which cause genital warts in some people. Gardasil has been approved by the Food and Drug Administration and is recommended for girls and women from ages 9-26 for the prevention of some types of cancer of the cervix, vagina and vulva as well as preventing some types of genital warts. In males that are 9-26 years old, the FDA has approved its use for prevention of some types of genital warts.

The Gardasil vaccine is made from a virus like particle and does not contain any live virus. Children with an allergy to yeast should not receive the vaccine since some components of the vaccine are made from yeast.

People who have undergone organ transplant are at increased risk of of developing genital warts and cancers related to HPV when compared to the general population. The American Society of Transplantation and the American Society of Transplant Surgeons recommend the vaccine for people with transplants.

Studies of other vaccines like Hepatitis B have shown children after transplant have less of a response to this vaccine and are not immune to the Hepatitis B virus. We are interested in seeing if your child will form antibodies (immune response) to the Gardasil vaccine.

Your child is being asked to be in the study because he or she is between the ages of 9-17 and has undergone a liver or kidney transplant more than 6 months ago and does not have any signs of organ rejection.

DETAILED DESCRIPTION:
Currently Merck manufactures the HPV (types 6, 11, 16, and 18) L1 virus like particle vaccine and a description has been reported previously. (18) Merck will supply the vaccine, which will be stored as directed by the manufacturer. The vaccine will be stored at the Medstar Research Institute (Women and Infants Research Services) It will be administered by intramuscular injection (0.5 mL) into the upper arm or thigh by the research nurse (Sarah Duwel, RN or a nurse working under supervision) in the transplant clinic.

Participants will be given a form to fill out regarding allergic prior to vaccination. After the research nurse reviews the form with the patient and their guardian, an immunization or blood collection will be performed. Participants will receive a full dose vaccine on day 1, at month 2 (± 3 weeks), and at month 6 (± 3 weeks). All participants will be required to be afebrile (oral temperature <37.8° C) within 24 hours before each injection.

All female participants will undergo urine pregnancy testing and will not be vaccinated if found to be pregnant. Female participants with a positive urine pregnancy test will be informed confidentially of their test results by the study nurse and will be referred to an OB/GYN for further care.

Serum samples will be obtained from all participants on day 1, at month 3, and at month 7. Samples will be de-identified and stored at -20°C or below and anti-HPV levels will be determined using an HPV type-specific competitive Luminex xMAP-based immunoassay (cLIA). (18) Merck will make arrangements for the labs tests. This assay measures only neutralizing anti-HPV antibodies, rather than the broad assortment of vaccine-induced anti-HPV antibodies. Antibody levels will be expressed as milliMerck units (mMU) per milliliter. The lower limits of detection for the anti-HPV 6, 11, 16, and 18 cLIAs are 4.1 mMU6/mL, 3.0 mMU11/mL, 10.2 mMU16/mL, and 2.9 mMU18/mL, respectively. Assay precision is estimated to be 21.7%, 20.4%, 23.0%, and 15.9% for the anti-HPV 6, 11, 16, and 18 cLIAs respectively. Participants will be considered anti-HPV 6, 11, 16, or 18 seropositive when their anti-HPV antibody titers are 20 mMU6/mL, 16 mMU11/mL, 20 mMU16/mL, or 24 mMU18/mL, respectively.

Blood collection supplies will be obtained from a lab vendor Laprepco (www.labrepco.com). The lab we will use to process our antibody titers is PPD Labs (www.ppdi.com). De-identified blood samples will be stored by the research nurse at Mesdstar Research Institute until they are able to be shipped to the PPD lab. Our research nurses are trained in Environmental and Health Safety training based on Medstar Research Institution requirements. Antibody titers results will be mail directly to Dr. Gomez-Lobo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 9-17 who have undergone liver or kidney transplant are on stable immunosuppressant doses for greater than 6 months

Exclusion Criteria:

* Previous vaccination with Gardasil or Cervarix
* Allergy to Gardasil or components of Gardasil including yeast
* Diagnosis of HIV or cancer
* Pregnancy
* Blood transfusion 6 months prior to initiation of Gardasil vaccine protocol

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2012-01-20 (Actual); Study Completion 2012-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Gomez-Lobo, MD, Principal Investigator — Washington Hospital Center, Georgetown University Hospital
Locations (2):
- United States (2):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Childrens National Medical Center, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Danzinger-Isakov L, Kumar D; AST Infectious Diseases Community of Practice. Guidelines for vaccination of solid organ transplant candidates and recipients. Am J Transplant. 2009 Dec;9 Suppl 4:S258-62. doi: 10.1111/j.1600-6143.2009.02917.x. No abstract available. PMID 20070687
- [Background] Kasiske BL, Snyder JJ, Gilbertson DT, Wang C. Cancer after kidney transplantation in the United States. Am J Transplant. 2004 Jun;4(6):905-13. doi: 10.1111/j.1600-6143.2004.00450.x. PMID 15147424
- [Background] De Vuyst H, Clifford GM, Nascimento MC, Madeleine MM, Franceschi S. Prevalence and type distribution of human papillomavirus in carcinoma and intraepithelial neoplasia of the vulva, vagina and anus: a meta-analysis. Int J Cancer. 2009 Apr 1;124(7):1626-36. doi: 10.1002/ijc.24116. PMID 19115209
- [Background] D'Souza G, Kreimer AR, Viscidi R, Pawlita M, Fakhry C, Koch WM, Westra WH, Gillison ML. Case-control study of human papillomavirus and oropharyngeal cancer. N Engl J Med. 2007 May 10;356(19):1944-56. doi: 10.1056/NEJMoa065497. PMID 17494927
- [Background] Badawi H, Ahmed H, Ismail A, Diab M, Moubarak M, Badawy A, Saber M. Role of human papillomavirus types 16, 18, and 52 in recurrent cystitis and urinary bladder cancer among Egyptian patients. Medscape J Med. 2008;10(10):232. Epub 2008 Oct 8. PMID 19099026
- [Background] Penn I. Occurrence of cancers in immunosuppressed organ transplant recipients. Clin Transpl. 1998:147-58. PMID 10503093
- [Background] Villa LL, Costa RL, Petta CA, Andrade RP, Paavonen J, Iversen OE, Olsson SE, Hoye J, Steinwall M, Riis-Johannessen G, Andersson-Ellstrom A, Elfgren K, Krogh Gv, Lehtinen M, Malm C, Tamms GM, Giacoletti K, Lupinacci L, Railkar R, Taddeo FJ, Bryan J, Esser MT, Sings HL, Saah AJ, Barr E. High sustained efficacy of a prophylactic quadrivalent human papillomavirus types 6/11/16/18 L1 virus-like particle vaccine through 5 years of follow-up. Br J Cancer. 2006 Dec 4;95(11):1459-66. doi: 10.1038/sj.bjc.6603469. Epub 2006 Nov 21. PMID 17117182
- [Background] Joura EA, Kjaer SK, Wheeler CM, Sigurdsson K, Iversen OE, Hernandez-Avila M, Perez G, Brown DR, Koutsky LA, Tay EH, Garcia P, Ault KA, Garland SM, Leodolter S, Olsson SE, Tang GW, Ferris DG, Paavonen J, Lehtinen M, Steben M, Bosch X, Dillner J, Kurman RJ, Majewski S, Munoz N, Myers ER, Villa LL, Taddeo FJ, Roberts C, Tadesse A, Bryan J, Lupinacci LC, Giacoletti KE, Lu S, Vuocolo S, Hesley TM, Haupt RM, Barr E. HPV antibody levels and clinical efficacy following administration of a prophylactic quadrivalent HPV vaccine. Vaccine. 2008 Dec 9;26(52):6844-51. doi: 10.1016/j.vaccine.2008.09.073. Epub 2008 Oct 16. PMID 18930097
- [Background] FUTURE II Study Group. Quadrivalent vaccine against human papillomavirus to prevent high-grade cervical lesions. N Engl J Med. 2007 May 10;356(19):1915-27. doi: 10.1056/NEJMoa061741. PMID 17494925
- [Background] Villa LL. Overview of the clinical development and results of a quadrivalent HPV (types 6, 11, 16, 18) vaccine. Int J Infect Dis. 2007 Nov;11 Suppl 2:S17-25. doi: 10.1016/S1201-9712(07)60017-4. PMID 18162241
- [Background] Carey W, Pimentel R, Westveer MK, Vogt D, Broughan T. Failure of hepatitis B immunization in liver transplant recipients: results of a prospective trial. Am J Gastroenterol. 1990 Dec;85(12):1590-2. PMID 2252022
- [Background] Guidelines for vaccination of solid organ transplant candidates and recipients. Am J Transplant. 2004 Nov;4 Suppl 10:160-3. doi: 10.1111/j.1600-6135.2004.00737.x. No abstract available. PMID 15504229
- [Background] Loinaz C, de Juanes JR, Gonzalez EM, Lopez A, Lumbreras C, Gomez R, Gonzalez-Pinto I, Jimenez C, Garcia I, Fuertes A. Hepatitis B vaccination results in 140 liver transplant recipients. Hepatogastroenterology. 1997 Jan-Feb;44(13):235-8. PMID 9058151
- [Background] Duca P, Del Pont JM, D'Agostino D. Successful immune response to a recombinant hepatitis B vaccine in children after liver transplantation. J Pediatr Gastroenterol Nutr. 2001 Feb;32(2):168-70. doi: 10.1097/00005176-200102000-00014. PMID 11321387
- [Background] Lefebure AF, Verpooten GA, Couttenye MM, De Broe ME. Immunogenicity of a recombinant DNA hepatitis B vaccine in renal transplant patients. Vaccine. 1993;11(4):397-9. doi: 10.1016/0264-410x(93)90278-6. PMID 8470423
- [Background] Rendi-Wagner P, Kundi M, Stemberger H, Wiedermann G, Holzmann H, Hofer M, Wiesinger K, Kollaritsch H. Antibody-response to three recombinant hepatitis B vaccines: comparative evaluation of multicenter travel-clinic based experience. Vaccine. 2001 Feb 28;19(15-16):2055-60. doi: 10.1016/s0264-410x(00)00410-2. PMID 11228377
- [Background] Block SL, Nolan T, Sattler C, Barr E, Giacoletti KE, Marchant CD, Castellsague X, Rusche SA, Lukac S, Bryan JT, Cavanaugh PF Jr, Reisinger KS; Protocol 016 Study Group. Comparison of the immunogenicity and reactogenicity of a prophylactic quadrivalent human papillomavirus (types 6, 11, 16, and 18) L1 virus-like particle vaccine in male and female adolescents and young adult women. Pediatrics. 2006 Nov;118(5):2135-45. doi: 10.1542/peds.2006-0461. PMID 17079588

RESULTS

PARTICIPANT FLOW:
Groups:
- Liver and Kidney Transplant Arm: Standard of Care Intervention: Participants on this arm receive Gardasil vaccine and have a history of liver or kidney transplant.
  Biological/Vaccine: Quadrivalent HPV for types 6, 11, 16 and 18 Per standard of care, Gardasil 0.5ml IM injection on day one, month 2, and month 6.
  Serum samples on day one, month 3 and month 7.
Period: Overall Study
Arm/Group | Liver and Kidney Transplant Arm
Started | 25
Completed | 9
Not Completed | 16

BASELINE CHARACTERISTICS:
Groups:
- Liver and Kidney Transplant Patient Arm: Standard of Care Intervention: Participants on this arm receive Gardasil vaccine and have a history of liver or kidney transplant.
  Biological/Vaccine: Quadrivalent HPV for types 6, 11, 16 and 18 Per standard of care, Gardasil 0.5ml IM injection on day one, month 2, and month 6.
  Serum samples on day one, month 3 and month 7.
Arm/Group | Liver and Kidney Transplant Patient Arm
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 15 [11 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 6
  More than one race | 7
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Showing Seroconversion to All HPV Four Serotypes
Time Frame: 7 months
Population: 9 of 25 patients completed the full study (three vaccinations and blood draws). Incomplete data was collected for the remaining 16 subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Liver and Kidney Transplant Patient Arm: Standard of Care Intervention: Participants on this arm receive Gardisil vaccine and have a history of liver transplant.
  Biological/Vaccine: Quadrivalent HPV for types 6, 11, 16 and 18 Per standard of care, Gardasil 0.5ml IM injection on day one, month 2, and month 6.
  Serum samples on day one, month 3 and month 7.
Arm/Group | Liver and Kidney Transplant Patient Arm
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Arm/Group | Liver and Kidney Transplant Arm
Serious Adverse Events (participants affected / at risk) | 3/25
Other Adverse Events (participants affected / at risk) | 9/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liver and Kidney Transplant Arm (N=25)
Acute graft rejection (Renal and urinary disorders) | 2 (2)
High grade fever (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liver and Kidney Transplant Arm (N=25)
Fever (Renal and urinary disorders) | 3
Facial Acne (Renal and urinary disorders) | 1
Swelling and Pain at the Injection Site (Renal and urinary disorders) | 3
Cough (Renal and urinary disorders) | 1
Pneumonia (Renal and urinary disorders) | 1
Diarrhea (Renal and urinary disorders) | 1
Headache (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes